CLINICAL TRIAL: NCT03433482
Title: Immunogenicity, Reactogenicity and Safety Study of Different Formulations of GSK Biologicals' Meningococcal ACWY Conjugate Vaccine (GSK3536820A and Menveo) When Administered to Healthy Adolescents and Young Adults 10 to 40 Years of Age
Brief Title: A Study to Investigate the Safety and Immunogenicity of Different Formulations of GSK Biologicals' Meningococcal ACWY Conjugate Vaccine (GSK3536820A and Menveo) Administered to Healthy Adolescents and Young Adults 10 to 40 Years of Age
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 207467; V59_78 (Other: Novartis); 2017-003456-23 (EudraCT Number)
Record Dates: First submitted 2018-02-08; First posted 2018-02-14 (Actual); Results first posted 2021-02-17 (Actual); Last update posted 2021-02-17 (Actual); Status verified 2021-01

CONDITIONS: Meningitis, Meningococcal
Keywords: Meningococcal disease; Liquid formulation; Meningitis
MeSH Terms: conditions — Meningitis, Meningococcal; Meningococcal Infections; Meningitis | interventions — MenACWY; Meningococcal Vaccines

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Data will be collected in an observer-blind manner. By observer-blind, it is meant that during the course of the study, the vaccine recipient and those responsible for the evaluation of any study endpoint (e.g. safety, reactogenicity and immunogenicity) will all be unaware of which vaccine was administered. To do so, vaccine preparation and administration will be done by authorized medical personnel who will not participate in any of the study clinical evaluations.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- GSK3536820A ACWY_Liq24 Group (Experimental): Healthy subjects receiving a single dose of the investigational MenACWY liquid vaccine formulation aged for approximately 24 months, at Day 1 in the Study Phase1.
  Interventions: Biological: MenACWY liquid
- ACWY_1 Group (Active Comparator): Healthy subjects receiving a single dose of the licensed GSK's MenACWY vaccine formulation (Menveo), at Day 1 in the Study Phase1.
  Interventions: Biological: MenACWY
- GSK3536820A ACWY_Liq30 Group (Experimental): Healthy subjects receiving a single dose of the investigational MenACWY liquid vaccine formulation aged for approximately 30 months, at Day 1 in the Study Phase 2.
  Interventions: Biological: MenACWY liquid
- ACWY_2 Group (Active Comparator): Healthy subjects receiving a single dose of the licensed GSK's MenACWY vaccine formulation (Menveo), at Day 1 in the Study Phase 2.
  Interventions: Biological: MenACWY

INTERVENTIONS:
Biological: MenACWY liquid — At visit 1 (day 1), each subject will receive a single dose of the investigational MenACWY liquid vaccine (GSK3536820A) aged for approximately 24 months in Phase 1 of the study (subjects randomized to study arm ACWY_Liq24) or vaccine aged for 30 months in Phase 2 of the study (subjects randomized to study arm ACWY_Liq30), administered by intramuscular injection in the deltoid of the non-dominant arm.
  Arms: GSK3536820A ACWY_Liq24 Group; GSK3536820A ACWY_Liq30 Group
Biological: MenACWY — At visit 1 (day 1), each subject will receive a single dose of the MenACWY vaccine in the Phase1 of the study (subjects randomized to study arm ACWY_1) or in phase 2 of the study (subjects randomized to study arm ACWY_2), administered by intramuscular injection in the deltoid of the non-dominant arm.
  Other Names: Menveo
  Arms: ACWY_1 Group; ACWY_2 Group

SUMMARY:
MenACWY (Menveo) is a GSK vaccine intended for protection against disease caused by meningococcal bacteria groups A, C, W and Y in infants, children and adults, licensed in more than 60 countries.

The purpose of this study is to compare the immunogenicity of the currently licensed MenACWY vaccine with the investigational MenACWY liquid vaccine aged for different lengths of time by storage at 2-8ºC.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects who, in the opinion of the investigator, can and will comply with the requirements of the protocol or subjects' parent(s)/Legally Acceptable Representative(s) [LAR(s)] who, in the opinion of the investigator, can and will comply, with the requirements of the protocol.
2. Written informed consent obtained from the subject/from the parent(s)/LAR(s) of the subject prior to performing any study specific procedure.
3. Written informed assent obtained for subjects below legal age of consent, if required by local regulations at the time of the enrolment.
4. A male or female ≥10 to ≤40 YoA at the time of the vaccination.
5. Healthy subjects as established by medical history and clinical examination before entering into the study.
6. Female subjects of non-childbearing potential may be enrolled in the study.

   * Non-childbearing potential is defined as pre-menarche, current bilateral tubal ligation or occlusion, hysterectomy, bilateral ovariectomy or post-menopause
7. Female subjects of childbearing potential may be enrolled in the study, if the subject:

   * has practiced adequate contraception for 30 days prior to vaccination, and
   * has a negative pregnancy test on the day of vaccination, and
   * has agreed to continue adequate contraception during the entire treatment period.

Exclusion Criteria:

1. Child in care
2. Anaphylaxis following the administration of vaccine.
3. Any (clinical) condition that in the judgment of the investigator would make intramuscular injection unsafe &/represents a contraindication to intramuscular vaccination and blood draws.
4. Any confirmed or suspected immunosuppressive or immunodeficient condition, including HIV infection.
5. Progressive, unstable or uncontrolled clinical conditions.
6. Hypersensitivity, including allergy, to any component of vaccines, medicinal products or medical equipment whose use is foreseen in this study.
7. Hypersensitivity to the active substances or to any of the excipients of the vaccine, including diphtheria toxoid (CRM197), or a life-threatening reaction after previous administration of a vaccine containing similar components.
8. Abnormal function of the immune system resulting from:

   * Clinical conditions.
   * Systemic administration of corticosteroids within 90 days prior to informed consent, and until the Day 29 blood draw.
   * Administration of antineoplastic and immunomodulating agents or radiotherapy within 90 days prior to informed consent, and until the Day 29 blood draw.
9. Received immunoglobulins or any blood products within 180 days prior to informed consent.
10. Received an investigational or non-registered medicinal product within 30 days prior to informed consent.
11. Any other clinical condition that, in the opinion of the investigator, might pose additional risk to the subject due to participation in the study.
12. History of any meningococcal vaccination, with the exception of previous meningococcal C vaccination, if the last dose of MenC was received at ≤24 months of age.
13. Individuals who received any other vaccines within 7 days (for inactivated vaccines) or 14 days prior to enrolment in this study or who are planning to receive any vaccine within 28 days from the study vaccines.*

    * In case an emergency mass vaccination for an unforeseen public health threat is organized by the public health authorities, outside the routine immunization program, the time period described above can be reduced if necessary for that vaccine provided it is licensed and used according to its Prescribing Information and according to the local governmental recommendations and provided a written approval of the sponsor is obtained.
14. Administration of long-acting immune-modifying drugs at any time during the study period (e.g. infliximab).
15. Concurrently participating in another clinical study, at any time during the study period, in which the subject has been or will be exposed to an investigational or a non-investigational vaccine/product (pharmaceutical product or device).
16. Current or previous, confirmed or suspected disease caused by N. meningitidis.
17. Household contact with and/or intimate exposure to an individual with any laboratory confirmed N. meningitidis infection within 60 days prior to study vaccination.
18. Acute disease and/or fever within 3 days prior to study vaccination. Note: enrolment may be postponed/delayed until such transient circumstances have ended.

    * Fever is defined as body temperature ≥38.0°C/100.4°F. The preferred location for measuring temperature in this study will be the oral cavity.
    * Subjects with a minor illness (such as mild diarrhoea, mild upper respiratory infection) without fever may be enrolled at the discretion of the investigator.
19. Received systemic antibiotic treatment within 3 days prior to study vaccination or blood draw.
20. Study personnel as an immediate family or household member.
21. Pregnant or lactating women.

Ages: 10 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 1707 (Actual)
Dates: Start 2018-08-30 (Actual); Primary Completion 2019-07-26 (Actual); Study Completion 2019-12-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (39):
- Brazil (4):
  - GSK Investigational Site, Salvador, Estado de Bahia
  - GSK Investigational Site, Natal, Rio Grande do Norte
  - GSK Investigational Site, Rio de Janeiro
  - GSK Investigational Site, São Paulo
- Estonia (2):
  - GSK Investigational Site, Tallinn
  - GSK Investigational Site, Tartu
- Finland (6):
  - GSK Investigational Site, Espoo
  - GSK Investigational Site, Helsinki
  - GSK Investigational Site, Jarvenpaa
  - GSK Investigational Site, Oulu
  - GSK Investigational Site, Pori
  - GSK Investigational Site, Tampere
- France (5):
  - GSK Investigational Site, Angers
  - GSK Investigational Site, Nantes
  - GSK Investigational Site, Nice
  - GSK Investigational Site, Rosiers-d'Égletons
  - GSK Investigational Site, Tours
- Mexico (2):
  - GSK Investigational Site, Mérida, Yucatán
  - GSK Investigational Site, Durango
- Russia (7):
  - GSK Investigational Site, Gatchina
  - GSK Investigational Site, Moscow
  - GSK Investigational Site, Murmansk
  - GSK Investigational Site, Saint Petersburg
  - GSK Investigational Site, Tomsk
  - GSK Investigational Site, Yaroslavl
  - GSK Investigational Site, Yekaterinburg
- South Africa (2):
  - GSK Investigational Site, Pretoria, Gauteng
  - GSK Investigational Site, Bellville
- Spain (9):
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, Centelles (Barcelona)
  - GSK Investigational Site, L'Hospitalet de Llobregat
  - GSK Investigational Site, La Roca Del Valles (Barcelona)
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Quart de Poblet, Valencia
  - GSK Investigational Site, Seville
  - GSK Investigational Site, Valencia
  - GSK Investigational Site, Vic/ Barcelona
- Turkey (Türkiye) (2):
  - GSK Investigational Site, Eskişehir
  - GSK Investigational Site, Izmir

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD will be made available within 6 months of publishing the results of the primary endpoints, key secondary endpoints and safety data of the study
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://clinicalstudydatarequest.com

REFERENCES:
- [Derived] Vir Singh P, Tiberi P, Di Domenico GF, Romolini V, Mzolo T, Costantini M, Akhund T, Basile V, Lattanzi M, Pellegrini M. Fully Liquid MenACWY-CRM Vaccine: Results from an Integrated Safety Analysis. Drug Saf. 2023 Jan;46(1):99-108. doi: 10.1007/s40264-022-01242-8. Epub 2022 Nov 11. PMID 36369456

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment was defined with 2 parallel groups per phase, in a 2-phase staggered design: Subjects in both experimental groups receiving investigational vaccine aged for approximately 24 months and 30 months in phase 1 and phase 2 respectively. Both comparator groups subjects in phase 1 and 2 of the study receiving licensed vaccine.
Pre-assignment Details: Out of the 1707 subjects enrolled in the study (inclusive of phase 1 and 2), 1690 were exposed to the vaccination. Out of the 17 subjects excluded from study, 11 were not randomized, 5 were not administered any study treatment, 1 did not sign the informed consent form.
Period: Overall Study
Arm/Group | GSK3536820A ACWY_Liq24 Group | ACWY_1 Group | GSK3536820A ACWY_Liq30 Group | ACWY_2 Group
Started | 420 | 424 | 427 | 419
Completed | 419 | 424 | 423 | 418
Not Completed | 1 | 0 | 4 | 1
Not completed — Lost to Follow-up | 1 | 0 | 1 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0
Not completed — Unknown reason | 0 | 0 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | GSK3536820A ACWY_Liq24 Group | ACWY_1 Group | GSK3536820A ACWY_Liq30 Group | ACWY_2 Group | Total
Number analyzed (Participants) | 420 | 424 | 427 | 419 | 1690
Age, Continuous [Mean (Standard Deviation); unit: Years] | 22.5 (9.4) | 22.2 (9.6) | 22.3 (9.8) | 22.0 (9.3) | 22.3 (9.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 232 | 242 | 259 | 228 | 961
  Male | 188 | 182 | 168 | 191 | 729
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian Or Alaska Native | 0 | 1 | 1 | 2 | 4
  Asian | 4 | 4 | 2 | 3 | 13
  Black Or African American | 26 | 22 | 30 | 26 | 104
  Other | 58 | 54 | 83 | 84 | 279
  White | 332 | 343 | 311 | 304 | 1290

OUTCOME MEASURES:

1. Primary Outcome: Adjusted Human Serum Bactericidal Activity (hSBA) Geometric Mean Titers (GMTs) Against N. Meningitidis Serogroup A for Each Vaccine Group and Between-group Ratios
Description: hSBA titers against N. meningitidis serogroup A are calculated in terms of GMTs adjusted for pre-vaccination titer.
Time Frame: At Day 29
Population: Analysis is performed on the per protocol set for immunogenicity that includes subjects who received the vaccine did not have any protocol deviation leading to exclusion , who were not excluded due to other reasons defined prior to unblinding or analysis and had available immuno data for any serogroup and time point considered.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | GSK3536820A ACWY_Liq24 Group | ACWY_1 Group | GSK3536820A ACWY_Liq30 Group | ACWY_2 Group
Number analyzed (Participants) | 363 | 373 | 356 | 349
Titers | 386.66 [319.47 to 467.97] | 318.34 [264.14 to 383.67] | 387.06 [322.72 to 464.24] | 348.89 [290.09 to 419.61]
Statistical Analysis 1: Comparison: GSK3536820A ACWY_Liq24 Group vs ACWY_1 Group; To demonstrate non-inferiority of the MenACWY liquid vaccine aged for approximately 24 months to that of currently licensed MenACWY vaccine, as measured by the adjusted hSBA GMTs directed against N. meningitidis serogroup A at Day 29 after a single dose vaccination; Test type: Non-Inferiority — Non-inferiority is concluded if the lower limit of the two sided 95% confidence interval (CI) for the hSBA GMT ratio for serogroup A between the MenACWY liquid vaccine aged for approximately 24 months and the licensed MenACWY vaccine is > 0.5; ANCOVA; Analysis of Covariance (ANCOVA) including pre-vaccination titer (Day 1) as a covariate and with vaccine group and country as factors; GMT ratio = 1.21, 95% CI 2-sided [0.94 to 1.57]
Statistical Analysis 2: Comparison: GSK3536820A ACWY_Liq30 Group vs ACWY_2 Group; To demonstrate non-inferiority of the MenACWY liquid vaccine aged for approximately 30 months to that of currently licensed MenACWY vaccine, as measured by the adjusted hSBA GMTs directed against N. meningitidis serogroup A at Day 29 after a single dose vaccination; Test type: Non-Inferiority — Non-inferiority is concluded if the lower limit of the two sided 95% CI for the hSBA GMT ratios for serogroup A between the MenACWY liquid vaccine aged for approximately 30 months and the licensed MenACWY vaccine is > 0.5. Non-inferiority hypotheses testing will be conducted sequentially, starting from MenACWY liquid vaccine aged for approximately 24 months and subsequently with MenACWY liquid vaccine aged for approximately 30 months; ANCOVA; [statistical method as in outcome 1, analysis 1]; GMT ratio = 1.11, 95% CI 2-sided [0.87 to 1.42]

2. Secondary Outcome: hSBA GMTs Against Each of the N.Meningitidis Serogroups A,C,W and Y for Each Vaccine Group and Between-group Ratios
Description: hSBA titers were calculated in terms of GMTs, at Day 1 and Day 29, against each of the N. meningitidis serogroup A, C, W and Y.
Time Frame: At Day 1 and Day 29
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | GSK3536820A ACWY_Liq24 Group | ACWY_1 Group | GSK3536820A ACWY_Liq30 Group | ACWY_2 Group
Number analyzed (Participants) | 394 | 398 | 395 | 392
Titers
  Meningitis A, Day 1: number analyzed (Participants) | 381 | 389 | 377 | 374
  Meningitis A, Day 1 | 3.01 [2.69 to 3.36] | 2.91 [2.60 to 3.24] | 3.34 [2.94 to 3.79] | 3.16 [2.78 to 3.59]
  Meningitis A, Day 29: number analyzed (Participants) | 363 | 373 | 356 | 349
  Meningitis A, Day 29 | 388.53 [320.61 to 470.84] | 319.06 [264.39 to 385.03] | 394.16 [326.72 to 475.50] | 349 [288.45 to 422.27]
  Meningitis C, Day 1: number analyzed (Participants) | 394 | 395 | 395 | 392
  Meningitis C, Day 1 | 8.59 [7.40 to 9.98] | 7.06 [6.09 to 8.20] | 9.05 [7.77 to 10.53] | 8.7 [7.46 to 10.14]
  Meningitis C, Day 29: number analyzed (Participants) | 385 | 377 | 376 | 377
  Meningitis C, Day 29 | 143.69 [109.13 to 189.20] | 157.74 [119.39 to 208.42] | 244.44 [182.20 to 327.96] | 208.34 [154.96 to 280.11]
  Meningitis W, Day 1: number analyzed (Participants) | 379 | 396 | 382 | 376
  Meningitis W, Day 1 | 6.23 [5.17 to 7.50] | 5.8 [4.83 to 6.95] | 5.69 [4.75 to 6.82] | 5.74 [4.78 to 6.90]
  Meningitis W, Day 29: number analyzed (Participants) | 372 | 388 | 374 | 366
  Meningitis W, Day 29 | 62.73 [49.93 to 78.81] | 63.92 [51.11 to 79.94] | 80.51 [64.66 to 100.24] | 73.08 [58.45 to 91.36]
  Meningitis Y, Day 1: number analyzed (Participants) | 390 | 398 | 391 | 385
  Meningitis Y, Day 1 | 4.39 [3.78 to 5.10] | 4.21 [3.63 to 4.89] | 4.14 [3.58 to 4.79] | 4.19 [3.62 to 4.86]
  Meningitis Y, Day 29: number analyzed (Participants) | 379 | 390 | 386 | 377
  Meningitis Y, Day 29 | 116.42 [94.03 to 144.15] | 105.11 [85.17 to 129.71] | 112.95 [91.55 to 139.34] | 118.04 [95.27 to 146.25]
Statistical Analysis 1: Comparison: GSK3536820A ACWY_Liq24 Group vs ACWY_1 Group; Between-groups ratio of adjusted hSBA GMTs and its 95% CI, between vaccine groups GSK3536820A ACWY_Liq24 and ACWY_1, at Day 29 against serogroup C; Test type: Other; ANCOVA; Analysis of Covariance (ANCOVA) including pre-vaccination titer (Day 1) as a covariate and with vaccine group and center (if applicable) as factors; GMT ratio = 0.84, 95% CI 2-sided [0.58 to 1.19]
Statistical Analysis 2: Comparison: GSK3536820A ACWY_Liq24 Group vs ACWY_1 Group; Between-groups ratio of adjusted hSBA GMTs and its 95% CI, between vaccine groups GSK3536820A ACWY_Liq24 and ACWY_1, at Day 29 against serogroup W; Test type: Other; ANCOVA; [statistical method as in outcome 2, analysis 1]; GMT ratio = 0.94, 95% CI 2-sided [0.72 to 1.24]
Statistical Analysis 3: Comparison: GSK3536820A ACWY_Liq24 Group vs ACWY_1 Group; Between-groups ratio of adjusted hSBA GMTs and its 95% CI, between vaccine groups GSK3536820A ACWY_Liq24 and ACWY_1, at Day 29 against serogroup Y; Test type: Other; ANCOVA; [statistical method as in outcome 2, analysis 1]; GMT ratio = 1.09, 95% CI 2-sided [0.82 to 1.44]
Statistical Analysis 4: Comparison: GSK3536820A ACWY_Liq30 Group vs ACWY_2 Group; Between-groups ratio of adjusted hSBA GMTs and its 95% CI, between vaccine groups GSK3536820A ACWY_Liq30 and ACWY_2, at Day 29 against serogroup C; Test type: Other; ANCOVA; [statistical method as in outcome 2, analysis 1]; GMT ratio = 1.14, 95% CI 2-sided [0.79 to 1.64]
Statistical Analysis 5: Comparison: GSK3536820A ACWY_Liq30 Group vs ACWY_2 Group; Between-groups ratio of adjusted hSBA GMTs and its 95% CI, between vaccine groups GSK3536820A ACWY_Liq30 and ACWY_2, at Day 29 against serogroup W; Test type: Other; ANCOVA; [statistical method as in outcome 2, analysis 1]; GMT ratio = 1.10, 95% CI 2-sided [0.84 to 1.45]
Statistical Analysis 6: Comparison: GSK3536820A ACWY_Liq30 Group vs ACWY_2 Group; Between-groups ratio of adjusted hSBA GMTs and its 95% CI, between vaccine groups GSK3536820A ACWY_Liq30 and ACWY_2, at Day 29 against serogroup Y; Test type: Other; ANCOVA; [statistical method as in outcome 2, analysis 1]; GMT ratio = 0.96, 95% CI 2-sided [0.72 to 1.26]

3. Secondary Outcome: Within-group Geometric Mean Ratios (GMRs) of GMTs Against Each of the N.Meningitidis Serogroups A,C,W and Y for Each Vaccine Group
Description: Within-group ratios of hSBA GMTs against each of the N.meningitidis serogroups A, C, W and Y at Day 29 compared to Day 1.
Time Frame: At Day 29
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | GSK3536820A ACWY_Liq24 Group | ACWY_1 Group | GSK3536820A ACWY_Liq30 Group | ACWY_2 Group
Number analyzed (Participants) | 385 | 390 | 386 | 377
Ratio
  Meningitis A: number analyzed (Participants) | 363 | 373 | 356 | 349
  Meningitis A | 130.33 [105.49 to 161.02] | 108.39 [88.14 to 133.30] | 114.66 [93.75 to 140.22] | 106.79 [87.05 to 131.01]
  Meningitis C: number analyzed (Participants) | 385 | 377 | 376 | 377
  Meningitis C | 17.01 [13.00 to 22.25] | 21.68 [16.52 to 28.46] | 26.69 [20.22 to 35.22] | 23.85 [18.04 to 31.54]
  Meningitis W: number analyzed (Participants) | 372 | 388 | 374 | 366
  Meningitis W | 9.81 [7.84 to 12.27] | 10.77 [8.65 to 13.41] | 13.8 [11.08 to 17.19] | 12.48 [9.98 to 15.61]
  Meningitis Y: number analyzed (Participants) | 379 | 390 | 386 | 377
  Meningitis Y | 26.53 [21.14 to 33.28] | 25.23 [20.18 to 31.54] | 27.18 [21.66 to 34.10] | 28.49 [22.60 to 35.92]

4. Secondary Outcome: Percentages of Subjects With ≥4 Fold Rise in hSBA Antibody Titers for Each of the N.Meningitidis Serogroups A, C,W and Y for Each Vaccine Group and Between-group Differences
Description: The percentages of subjects with a ≥ 4-fold rise in post-vaccination hSBA (at Day 29 compared to Day 1) and associated 2-sided 95% Clopper-Pearson CIs are computed by group and N. meningitidis serogroups A, C, W and Y. A 4-fold rise in the hSBA titers is defined as: - for individuals, whose pre-vaccination titers are < the LOD (limit of detection), the post-vaccination titers must be ≥ 4-fold the LOD or ≥ the LLOQ (lower limit of quantitation) whichever is greater; - for individuals whose pre-vaccination titers are ≥ the LOD and ≤ the LLOQ, the post-vaccination titers must be at least four times the LLOQ; - for individuals whose pre-vaccination titers are > the LLOQ, the post-vaccination titers must be at least four times the pre-vaccination titer.
Time Frame: At Day 29
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | GSK3536820A ACWY_Liq24 Group | ACWY_1 Group | GSK3536820A ACWY_Liq30 Group | ACWY_2 Group
Number analyzed (Participants) | 385 | 390 | 386 | 377
Percentage of subjects
  Meningitis A: number analyzed (Participants) | 363 | 373 | 356 | 349
  Meningitis A | 92.29 [89.04 to 94.81] | 90.08 [86.59 to 92.92] | 91.57 [88.19 to 94.24] | 91.69 [88.28 to 94.36]
  Meningitis C: number analyzed (Participants) | 385 | 377 | 376 | 377
  Meningitis C | 62.34 [57.29 to 67.20] | 64.46 [59.39 to 69.29] | 72.61 [67.80 to 77.05] | 69.76 [64.85 to 74.36]
  Meningitis W: number analyzed (Participants) | 372 | 388 | 374 | 366
  Meningitis W | 59.41 [54.23 to 64.44] | 60.57 [55.51 to 65.46] | 66.58 [61.55 to 71.34] | 62.57 [57.39 to 67.54]
  Meningitis Y: number analyzed (Participants) | 379 | 390 | 386 | 377
  Meningitis Y | 71.77 [66.95 to 76.25] | 73.33 [68.65 to 77.66] | 74.35 [69.69 to 78.64] | 77.19 [72.62 to 81.33]
Statistical Analysis 1: Comparison: GSK3536820A ACWY_Liq24 Group vs ACWY_1 Group; Between-group difference in percentage of subjects with a ≥ 4-fold rise in post-vaccination hSBA for N. meningitidis serogroup A at Day 29; Test type: Other; Miettinen and Nurminen score method; Difference in percentage of subjects = 2.21, 95% CI 2-sided [-1.94 to 6.40]
Statistical Analysis 2: Comparison: GSK3536820A ACWY_Liq24 Group vs ACWY_1 Group; Between-group difference in percentage of subjects with a ≥ 4-fold rise in post-vaccination hSBA for N. meningitidis serogroup C at Day 29; Test type: Other; Miettinen and Nurminen score method; Difference in percentage of subjects = -2.12, 95% CI 2-sided [-8.94 to 4.72]
Statistical Analysis 3: Comparison: GSK3536820A ACWY_Liq24 Group vs ACWY_1 Group; Between-group difference in percentage of subjects with a ≥ 4-fold rise in post-vaccination hSBA for N. meningitidis serogroup W at Day 29; Test type: Other; Miettinen and Nurminen score method; Difference in percentage of subjects = -1.16, 95% CI 2-sided [-8.11 to 5.80]
Statistical Analysis 4: Comparison: GSK3536820A ACWY_Liq24 Group vs ACWY_1 Group; Between-group difference in percentage of subjects with a ≥ 4-fold rise in post-vaccination hSBA for N. meningitidis serogroup Y at Day 29; Test type: Other; Miettinen and Nurminen score method; Difference in percentage of subjects = -1.57, 95% CI 2-sided [-7.88 to 4.74]
Statistical Analysis 5: Comparison: GSK3536820A ACWY_Liq30 Group vs ACWY_2 Group; [analysis description as in outcome 4, analysis 1]; Test type: Other; Miettinen and Nurminen score method; Difference in percentage of subjects = -0.12, 95% CI 2-sided [-4.29 to 4.07]
Statistical Analysis 6: Comparison: GSK3536820A ACWY_Liq30 Group vs ACWY_2 Group; [analysis description as in outcome 4, analysis 2]; Test type: Other; Miettinen and Nurminen score method; Difference in percentage of subjects = 2.85, 95% CI 2-sided [-3.63 to 9.30]
Statistical Analysis 7: Comparison: GSK3536820A ACWY_Liq30 Group vs ACWY_2 Group; [analysis description as in outcome 4, analysis 3]; Test type: Other; Miettinen and Nurminen score method; Difference in percentage of subjects = 4.01, 95% CI 2-sided [-2.89 to 10.88]
Statistical Analysis 8: Comparison: GSK3536820A ACWY_Liq30 Group vs ACWY_2 Group; [analysis description as in outcome 4, analysis 4]; Test type: Other; Miettinen and Nurminen score method; Difference in percentage of subjects = -2.84, 95% CI 2-sided [-8.91 to 3.26]

5. Secondary Outcome: Percentages of Subjects With hSBA Antibody Titers ≥8 Against Each of the N.Meningitidis Serogroups A,C,W and Y for Each Vaccine Group and Between-group Differences
Description: For each vaccine group the percentage of subjects with hSBA titer ≥8 , and its associated two-sided 95% Clopper-Pearson CIs are computed for each of the N. meningitidis serogroups A, C, W and Y.
Time Frame: At Day 1 and Day 29
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | GSK3536820A ACWY_Liq24 Group | ACWY_1 Group | GSK3536820A ACWY_Liq30 Group | ACWY_2 Group
Number analyzed (Participants) | 394 | 398 | 395 | 392
Percentage of subjects
  Meningitis A, Day 1: number analyzed (Participants) | 381 | 389 | 377 | 374
  Meningitis A, Day 1 | 12.07 [8.98 to 15.77] | 10.28 [7.45 to 13.74] | 13.53 [10.24 to 17.40] | 12.03 [8.91 to 15.77]
  Meningitis A, Day 29: number analyzed (Participants) | 378 | 384 | 377 | 367
  Meningitis A, Day 29 | 93.65 [90.70 to 95.89] | 92.19 [89.03 to 94.67] | 93.37 [90.37 to 95.66] | 94.01 [91.06 to 96.21]
  Meningitis C, Day 1: number analyzed (Participants) | 394 | 395 | 395 | 392
  Meningitis C, Day 1 | 48.48 [43.44 to 53.53] | 41.52 [36.61 to 46.55] | 50.63 [45.59 to 55.67] | 50.26 [45.19 to 55.31]
  Meningitis C, Day 29: number analyzed (Participants) | 388 | 382 | 379 | 379
  Meningitis C, Day 29 | 77.58 [73.10 to 81.63] | 78.01 [73.52 to 82.06] | 84.17 [80.10 to 87.70] | 82.85 [78.67 to 86.51]
  Meningitis W, Day 1: number analyzed (Participants) | 379 | 396 | 382 | 376
  Meningitis W, Day 1 | 31.66 [27.01 to 36.61] | 28.54 [24.14 to 33.26] | 28.8 [24.30 to 33.62] | 30.05 [25.46 to 34.96]
  Meningitis W, Day 29: number analyzed (Participants) | 389 | 392 | 389 | 384
  Meningitis W, Day 29 | 79.43 [75.07 to 83.34] | 80.87 [76.62 to 84.64] | 85.86 [82.00 to 89.17] | 81.77 [77.54 to 85.50]
  Meningitis Y, Day 1: number analyzed (Participants) | 390 | 398 | 391 | 385
  Meningitis Y, Day 1 | 22.82 [18.75 to 27.31] | 21.86 [17.90 to 26.25] | 21.48 [17.51 to 25.89] | 22.34 [18.27 to 26.83]
  Meningitis Y, Day 29: number analyzed (Participants) | 384 | 392 | 393 | 386
  Meningitis Y, Day 29 | 87.5 [83.77 to 90.64] | 85.46 [81.57 to 88.80] | 88.04 [84.42 to 91.08] | 87.56 [83.85 to 90.69]
Statistical Analysis 1: Comparison: GSK3536820A ACWY_Liq24 Group vs ACWY_1 Group; Between-group difference in percentages of subjects with hSBA titer ≥8 for the N. meningitidis serogroup A on Day 1; Test type: Other; Miettinen and Nurminen score method; Difference in percentage of subjects = 1.79, 95% CI 2-sided [-2.69 to 6.32]
Statistical Analysis 2: Comparison: GSK3536820A ACWY_Liq24 Group vs ACWY_1 Group; Between-group difference in percentages of subjects with hSBA titer ≥8 for the N. meningitidis serogroup C on Day 1; Test type: Other; Miettinen and Nurminen score method; Difference in percentage of subjects = 6.96, 95% CI 2-sided [0.01 to 13.84]
Statistical Analysis 3: Comparison: GSK3536820A ACWY_Liq24 Group vs ACWY_1 Group; Between-group difference in percentages of subjects with hSBA titer ≥8 for the N. meningitidis serogroup W on Day 1; Test type: Other; Miettinen and Nurminen score method; Difference in percentage of subjects = 3.13, 95% CI 2-sided [-3.33 to 9.58]
Statistical Analysis 4: Comparison: GSK3536820A ACWY_Liq24 Group vs ACWY_1 Group; Between-group difference in percentages of subjects with hSBA titer ≥8 for the N. meningitidis serogroup Y on Day 1; Test type: Other; Miettinen and Nurminen score method; Difference in percentage of subjects = 0.96, 95% CI 2-sided [-4.86 to 6.80]
Statistical Analysis 5: Comparison: GSK3536820A ACWY_Liq24 Group vs ACWY_1 Group; Between-group difference in percentages of subjects with hSBA titer ≥8 for the N. meningitidis serogroup A on Day 29; Test type: Other; Miettinen and Nurminen score method; Difference in percentage of subjects = 1.46, 95% CI 2-sided [-2.24 to 5.22]
Statistical Analysis 6: Comparison: GSK3536820A ACWY_Liq24 Group vs ACWY_1 Group; Between-group difference in percentages of subjects with hSBA titer ≥8 for the N. meningitidis serogroup C on Day 29; Test type: Other; Miettinen and Nurminen score method; Difference in percentage of subjects = -0.43, 95% CI 2-sided [-6.32 to 5.46]
Statistical Analysis 7: Comparison: GSK3536820A ACWY_Liq24 Group vs ACWY_1 Group; Between-group difference in percentages of subjects with hSBA titer ≥8 for the N. meningitidis serogroup W on Day 29; Test type: Other; Miettinen and Nurminen score method; Difference in percentage of subjects = -1.43, 95% CI 2-sided [-7.05 to 4.18]
Statistical Analysis 8: Comparison: GSK3536820A ACWY_Liq24 Group vs ACWY_1 Group; Between-group difference in percentages of subjects with hSBA titer ≥8 for the N. meningitidis serogroup Y on Day 29; Test type: Other; Miettinen and Nurminen score method; Difference in percentage of subjects = 2.04, 95% CI 2-sided [-2.81 to 6.90]
Statistical Analysis 9: Comparison: GSK3536820A ACWY_Liq30 Group vs ACWY_2 Group; Between-group difference in percentages of subjects with hSBA titer ≥8 for the N. meningitidis serogroup A on Day 1; Test type: Other; Miettinen and Nurminen score method; Difference in percentage of subjects = 1.50, 95% CI 2-sided [-3.32 to 6.33]
Statistical Analysis 10: Comparison: GSK3536820A ACWY_Liq30 Group vs ACWY_2 Group; Between-group difference in percentages of subjects with hSBA titer ≥8 for the N. meningitidis serogroup C on Day 1; Test type: Other; Miettinen and Nurminen score method; Difference in percentage of subjects = 0.38, 95% CI 2-sided [-6.60 to 7.35]
Statistical Analysis 11: Comparison: GSK3536820A ACWY_Liq30 Group vs ACWY_2 Group; Between-group difference in percentages of subjects with hSBA titer ≥8 for the N. meningitidis serogroup W on Day 1; Test type: Other; Miettinen and Nurminen score method; Difference in percentage of subjects = -1.26, 95% CI 2-sided [-7.75 to 5.23]
Statistical Analysis 12: Comparison: GSK3536820A ACWY_Liq30 Group vs ACWY_2 Group; Between-group difference in percentages of subjects with hSBA titer ≥8 for the N. meningitidis serogroup Y on Day 1; Test type: Other; Miettinen and Nurminen score method; Difference in percentage of subjects = -0.85, 95% CI 2-sided [-6.69 to 4.98]
Statistical Analysis 13: Comparison: GSK3536820A ACWY_Liq30 Group vs ACWY_2 Group; Between-group difference in percentages of subjects with hSBA titer ≥8 for the N. meningitidis serogroup A on Day 29; Test type: Other; Miettinen and Nurminen score method; Difference in percentage of subjects = -0.64, 95% CI 2-sided [-4.24 to 2.96]
Statistical Analysis 14: Comparison: GSK3536820A ACWY_Liq30 Group vs ACWY_2 Group; Between-group difference in percentages of subjects with hSBA titer ≥8 for the N. meningitidis serogroup C on Day 29; Test type: Other; Miettinen and Nurminen score method; Difference in percentage of subjects = 1.32, 95% CI 2-sided [-3.99 to 6.64]
Statistical Analysis 15: Comparison: GSK3536820A ACWY_Liq30 Group vs ACWY_2 Group; Between-group difference in percentages of subjects with hSBA titer ≥8 the N. meningitidis serogroup W on Day 29; Test type: Other; Miettinen and Nurminen score method; Difference in percentage of subjects = 4.09, 95% CI 2-sided [-1.11 to 9.33]
Statistical Analysis 16: Comparison: GSK3536820A ACWY_Liq30 Group vs ACWY_2 Group; Between-group difference in percentages of subjects with hSBA titer ≥8 for the N. meningitidis serogroup Y on Day 29; Test type: Other; Miettinen and Nurminen score method; Difference in percentage of subjects = 0.48, 95% CI 2-sided [-4.16 to 5.13]

6. Secondary Outcome: Percentages of Subjects With hSBA Titers ≥LLOQ Against Each of the N. Meningitidis Serogroups A, C, W and Y for Each Vaccine Group, and Between-group Differences
Description: For each vaccine group the percentages of subjects with hSBA titer ≥LLOQ, and its associated two-sided 95% Clopper-Pearson CIs are computed for each of the N. meningitidis serogroups A, C, W and Y.
Time Frame: At Day 1 and Day 29
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | GSK3536820A ACWY_Liq24 Group | ACWY_1 Group | GSK3536820A ACWY_Liq30 Group | ACWY_2 Group
Number analyzed (Participants) | 394 | 398 | 395 | 392
Percentage of subjects
  Meningitis A, Day 1: number analyzed (Participants) | 381 | 389 | 377 | 374
  Meningitis A, Day 1 | 12.86 [9.67 to 16.64] | 11.57 [8.56 to 15.17] | 15.38 [11.89 to 19.43] | 13.64 [10.32 to 17.54]
  Meningitis A, Day 29: number analyzed (Participants) | 378 | 384 | 377 | 367
  Meningitis A, Day 29 | 93.92 [91.01 to 96.10] | 92.19 [89.03 to 94.67] | 93.37 [90.37 to 95.66] | 94.01 [91.06 to 96.21]
  Meningitis C, Day 1: number analyzed (Participants) | 394 | 395 | 395 | 392
  Meningitis C, Day 1 | 55.84 [50.78 to 60.81] | 48.61 [43.58 to 53.66] | 61.01 [56.01 to 65.85] | 57.14 [52.08 to 62.10]
  Meningitis C, Day 29: number analyzed (Participants) | 388 | 382 | 379 | 379
  Meningitis C, Day 29 | 79.38 [75.01 to 83.30] | 80.37 [76.02 to 84.23] | 84.7 [80.67 to 88.17] | 84.7 [80.67 to 88.17]
  Meningitis W, Day 1: number analyzed (Participants) | 379 | 396 | 382 | 376
  Meningitis W, Day 1 | 32.45 [27.76 to 37.42] | 28.54 [24.14 to 33.26] | 29.32 [24.80 to 34.16] | 30.05 [25.46 to 34.96]
  Meningitis W, Day 29: number analyzed (Participants) | 389 | 392 | 389 | 384
  Meningitis W, Day 29 | 79.43 [75.07 to 83.34] | 80.87 [76.62 to 84.64] | 85.86 [82.00 to 89.17] | 81.77 [77.54 to 85.50]
  Meningitis Y, Day 1: number analyzed (Participants) | 390 | 398 | 391 | 385
  Meningitis Y, Day 1 | 24.36 [20.18 to 28.93] | 22.86 [18.83 to 27.31] | 21.74 [17.75 to 26.16] | 22.86 [18.76 to 27.38]
  Meningitis Y, Day 29: number analyzed (Participants) | 384 | 392 | 393 | 386
  Meningitis Y, Day 29 | 88.28 [84.63 to 91.32] | 86.22 [82.41 to 89.48] | 88.3 [84.70 to 91.30] | 87.56 [83.85 to 90.69]
Statistical Analysis 1: Comparison: GSK3536820A ACWY_Liq24 Group vs ACWY_1 Group; Between-group difference in percentages of subjects with hSBA titer ≥LLOQ for the N. meningitidis serogroup A at Day 1; Test type: Other; Miettinen and Nurminen score method; Difference in percentage of subjects = 1.29, 95% CI 2-sided [-3.37 to 5.99]
Statistical Analysis 2: Comparison: GSK3536820A ACWY_Liq24 Group vs ACWY_1 Group; Between-group difference in percentages of subjects with hSBA titer ≥LLOQ for the N. meningitidis serogroup C at Day 1; Test type: Other; Miettinen and Nurminen score method; Difference in percentage of subjects = 7.23, 95% CI 2-sided [0.25 to 14.13]
Statistical Analysis 3: Comparison: GSK3536820A ACWY_Liq24 Group vs ACWY_1 Group; Between-group difference in percentages of subjects with hSBA titer ≥LLOQ for the N. meningitidis serogroup W at Day 1; Test type: Other; Miettinen and Nurminen score method; Difference in percentage of subjects = 3.92, 95% CI 2-sided [-2.57 to 10.39]
Statistical Analysis 4: Comparison: GSK3536820A ACWY_Liq24 Group vs ACWY_1 Group; Between-group difference in percentages of subjects with hSBA titer ≥LLOQ for the N. meningitidis serogroup Y at Day 1; Test type: Other; Miettinen and Nurminen score method; Difference in percentage of subjects = 1.49, 95% CI 2-sided [-4.44 to 7.44]
Statistical Analysis 5: Comparison: GSK3536820A ACWY_Liq24 Group vs ACWY_1 Group; Between-group difference in percentages of subjects with hSBA titer ≥LLOQ for the N. meningitidis serogroup A at Day 29; Test type: Other; Miettinen and Nurminen score method; Difference in percentage of subjects = 1.73, 95% CI 2-sided [-1.94 to 5.46]
Statistical Analysis 6: Comparison: GSK3536820A ACWY_Liq24 Group vs ACWY_1 Group; Between-group difference in percentages of subjects with hSBA titer ≥LLOQ for the N. meningitidis serogroup C at Day 29; Test type: Other; Miettinen and Nurminen score method; Difference in percentage of subjects = -0.99, 95% CI 2-sided [-6.66 to 4.70]
Statistical Analysis 7: Comparison: GSK3536820A ACWY_Liq24 Group vs ACWY_1 Group; Between-group difference in percentages of subjects with hSBA titer ≥LLOQ for the N. meningitidis serogroup W at Day 29; Test type: Other; Miettinen and Nurminen score method; Difference in percentage of subjects = -1.43, 95% CI 2-sided [-7.05 to 4.18]
Statistical Analysis 8: Comparison: GSK3536820A ACWY_Liq24 Group vs ACWY_1 Group; Between-group difference in percentages of subjects with hSBA titer ≥LLOQ for the N. meningitidis serogroup Y at Day 29; Test type: Other; Miettinen and Nurminen score method; Difference in percentage of subjects = 2.06, 95% CI 2-sided [-2.67 to 6.80]
Statistical Analysis 9: Comparison: GSK3536820A ACWY_Liq30 Group vs ACWY_2 Group; Between-group difference in percentages of subjects with hSBA titer ≥LLOQ for the N. meningitidis serogroup A at Day 1; Test type: Other; Miettinen and Nurminen score method; Difference in percentage of subjects = 1.75, 95% CI 2-sided [-3.32 to 6.83]
Statistical Analysis 10: Comparison: GSK3536820A ACWY_Liq30 Group vs ACWY_2 Group; Between-group difference in percentages of subjects with hSBA titer ≥LLOQ for the N. meningitidis serogroup C at Day 1; Test type: Other; Miettinen and Nurminen score method; Difference in percentage of subjects = 3.87, 95% CI 2-sided [-3.00 to 10.71]
Statistical Analysis 11: Comparison: GSK3536820A ACWY_Liq30 Group vs ACWY_2 Group; Between-group difference in percentages of subjects with hSBA titer ≥LLOQ for the N. meningitidis serogroup W at Day 1; Test type: Other; Miettinen and Nurminen score method; Difference in percentage of subjects = -0.73, 95% CI 2-sided [-7.24 to 5.77]
Statistical Analysis 12: Comparison: GSK3536820A ACWY_Liq30 Group vs ACWY_2 Group; Between-group difference in percentages of subjects with hSBA titer ≥LLOQ for the N. meningitidis serogroup Y at Day 1; Test type: Other; Miettinen and Nurminen score method; Difference in percentage of subjects = -1.12, 95% CI 2-sided [-6.99 to 4.75]
Statistical Analysis 13: Comparison: GSK3536820A ACWY_Liq30 Group vs ACWY_2 Group; Between-group difference in percentages of subjects with hSBA titer ≥LLOQ for the N. meningitidis serogroup A at Day 29; Test type: Other; Miettinen and Nurminen score method; Difference in percentage of subjects = -0.64, 95% CI 2-sided [-4.24 to 2.96]
Statistical Analysis 14: Comparison: GSK3536820A ACWY_Liq30 Group vs ACWY_2 Group; Between-group difference in percentages of subjects with hSBA titer ≥LLOQ for the N. meningitidis serogroup C at Day 29; Test type: Other; Miettinen and Nurminen score method; Difference in percentage of subjects = 0.00, 95% CI 2-sided [-5.16 to 5.16]
Statistical Analysis 15: Comparison: GSK3536820A ACWY_Liq30 Group vs ACWY_2 Group; Between-group difference in percentages of subjects with hSBA titer ≥LLOQ for the N. meningitidis serogroup W at Day 29; Test type: Other; Miettinen and Nurminen score method; Difference in percentage of subjects = 4.09, 95% CI 2-sided [-1.11 to 9.33]
Statistical Analysis 16: Comparison: GSK3536820A ACWY_Liq30 Group vs ACWY_2 Group; Between-group difference in percentages of subjects with hSBA titer ≥LLOQ for the N. meningitidis serogroup Y at Day 29; Test type: Other; Miettinen and Nurminen score method; Difference in percentage of subjects = 0.73, 95% CI 2-sided [-3.88 to 5.37]

7. Secondary Outcome: Number of Subjects Reported With Any Unsolicited Adverse Events (AEs) Within 30 Minutes After Vaccination
Description: An unsolicited adverse event (AE) is defined as any untoward medical occurrence in a subject or clinical investigation subject administered with a pharmaceutical product at any dose that does not necessarily have to have a causal relationship with this treatment.
Time Frame: Within 30 minutes after vaccination at Day 1
Population: Analysis was performed on the unsolicited safety set that includes all enrolled subjects who received a study vaccination and reported unsolicited adverse events data for the defined period.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK3536820A ACWY_Liq24 Group | ACWY_1 Group | GSK3536820A ACWY_Liq30 Group | ACWY_2 Group
Number analyzed (Participants) | 420 | 424 | 427 | 419
Participants | 2 | 2 | 6 | 6

8. Secondary Outcome: Number of Subjects Reported With Solicited Local and Systemic AEs
Description: Assessed solicited local AEs were erythema, induration and pain at injection site. Assessed solicited systemic AEs were Arthralgia, chills, fatigue, fever (body temperature ≥38.0°C), headache, loss of appetite, myalgia and nausea.
Time Frame: From Day 1 (6 hours) to Day 7 after vaccination
Population: Analysis was performed on the solicited safety set that includes all enrolled subjects who received a study vaccination and reported solicited adverse events data for the defined period.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK3536820A ACWY_Liq24 Group | ACWY_1 Group | GSK3536820A ACWY_Liq30 Group | ACWY_2 Group
Number analyzed (Participants) | 418 | 422 | 425 | 419
Participants
  Arthralgia | 45 | 50 | 49 | 40
  Chills | 75 | 79 | 78 | 56
  Erythema | 48 | 51 | 58 | 40
  Fatigue | 174 | 175 | 149 | 147
  Fever (Temperature >= 38 C) | 15 | 18 | 15 | 12
  Headache | 164 | 151 | 169 | 157
  Induration | 50 | 51 | 54 | 39
  Loss of Appetite | 53 | 54 | 63 | 34
  Myalgia | 60 | 59 | 58 | 65
  Nausea | 54 | 48 | 42 | 46
  Pain | 189 | 181 | 202 | 192

9. Secondary Outcome: Number of Subjects Reported With Other Indicators of Reactogenicity
Description: Number of subjects reporting other indicators of reactogenicity such as use of analgesics/antipyretics within 7 days after any vaccination
Time Frame: From Day 1 to Day 7 after vaccination
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | GSK3536820A ACWY_Liq24 Group | ACWY_1 Group | GSK3536820A ACWY_Liq30 Group | ACWY_2 Group
Number analyzed (Participants) | 418 | 422 | 425 | 419
Participants
  Analgesic/Antipyretic Prevention, No | 357 | 374 | 366 | 369
  Analgesic/Antipyretic Prevention, Yes | 61 | 48 | 59 | 50
  Analgesic/Antipyretic Treatment, No | 328 | 340 | 349 | 350
  Analgesic/Antipyretic Treatment, Yes | 90 | 82 | 76 | 69

10. Secondary Outcome: Number of Subjects Reported With Any Unsolicited AEs Within 29 Days After Vaccination
Description: as for outcome 7
Time Frame: From Day 1 to Day 29 after vaccination
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | GSK3536820A ACWY_Liq24 Group | ACWY_1 Group | GSK3536820A ACWY_Liq30 Group | ACWY_2 Group
Number analyzed (Participants) | 420 | 424 | 427 | 419
Participants | 77 | 91 | 101 | 97

11. Secondary Outcome: Number of Subjects Reported With Serious Adverse Events (SAEs), AEs Leading to Withdrawal and Medically Attended AEs
Description: Medically attended AEs are defined as events for which the subject received medical attention defined as hospitalization, an emergency room visit, or a visit to or from medical personnel (medical doctor) for any reason. Any medically attended AE(s) is occurrence of any medically attended AE(s) regardless of intensity grade or relation to vaccination. Serious adverse event is any congenital anomaly/birth defect in the offspring of a study subject or any untoward medical occurrence that results in death or life threatening or requires hospitalization or results in disability or incapacity
Time Frame: From Day 1 to Day 181 (during the entire study period)
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | GSK3536820A ACWY_Liq24 Group | ACWY_1 Group | GSK3536820A ACWY_Liq30 Group | ACWY_2 Group
Number analyzed (Participants) | 420 | 424 | 427 | 419
Participants
  AEs Leading to withdrawal | 0 | 0 | 0 | 0
  SAEs | 4 | 1 | 4 | 4
  Medically attended AEs | 88 | 69 | 81 | 77

ADVERSE EVENTS:
Time Frame: Solicited AEs were collected from Day 1 to Day 7 after vaccination and Unsolicited AEs from Day 1 to Day 29 after vaccination. SAEs were collected from Day 1 to Day 181 (during the entire study period)
Arm/Group | GSK3536820A ACWY_Liq24 Group | ACWY_1 Group | GSK3536820A ACWY_Liq30 Group | ACWY_2 Group
All-Cause Mortality (participants affected / at risk) | 0/420 | 0/424 | 0/427 | 0/419
Serious Adverse Events (participants affected / at risk) | 4/420 | 1/424 | 4/427 | 4/419
Other Adverse Events (participants affected / at risk) | 312/420 | 314/424 | 324/427 | 317/419
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GSK3536820A ACWY_Liq24 Group (N=420) | ACWY_1 Group (N=424) | GSK3536820A ACWY_Liq30 Group (N=427) | ACWY_2 Group (N=419)
Phimosis (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Appendicitis noninfective (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Otitis externa (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tooth abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Soft tissue injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tibia fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tension headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Adnexa uteri pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ovarian cyst ruptured (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GSK3536820A ACWY_Liq24 Group (N=420) | ACWY_1 Group (N=424) | GSK3536820A ACWY_Liq30 Group (N=427) | ACWY_2 Group (N=419)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Eye paraesthesia (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vision blurred (Eye disorders) | 1 (2) | 0 (0) | 0 (0) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 4 (4) | 4 (4) | 4 (4) | 6 (7)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dental caries (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 3 (4) | 0 (0) | 6 (6) | 5 (5)
Enteritis (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 54 (56) | 48 (49) | 43 (45) | 46 (46)
Odynophagia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Oesophagitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Toothache (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Administration site erythema (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Administration site induration (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Administration site pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Application site erythema (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Application site warmth (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chills (General disorders) | 77 (78) | 79 (81) | 78 (78) | 56 (57)
Discomfort (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Facial pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 175 (175) | 175 (179) | 150 (157) | 147 (150)
Induration (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Injection site erythema (General disorders) | 50 (51) | 51 (52) | 59 (68) | 42 (47)
Injection site haematoma (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Injection site induration (General disorders) | 52 (53) | 51 (51) | 54 (62) | 39 (43)
Injection site oedema (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Injection site pain (General disorders) | 190 (193) | 182 (183) | 205 (214) | 194 (201)
Injection site pruritus (General disorders) | 2 (3) | 3 (3) | 2 (2) | 2 (2)
Injection site rash (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Injection site scab (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Malaise (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Oedema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pain (General disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Pyrexia (General disorders) | 20 (21) | 19 (20) | 19 (19) | 14 (14)
Vaccination site pain (General disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Vessel puncture site induration (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vessel puncture site pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Allergy to arthropod sting (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Drug hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abscess limb (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abscess oral (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acute sinusitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Balanitis candida (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 0 (0) | 3 (3) | 0 (0) | 1 (1)
Conjunctivitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Enterobiasis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Helicobacter infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Herpes simplex (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Hordeolum (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 1 (1) | 2 (2) | 3 (3) | 3 (3)
Injection site cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Laryngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 7 (7) | 15 (15) | 6 (7) | 6 (6)
Oral candidiasis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oral herpes (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Otitis media (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Paronychia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 2 (3) | 1 (1)
Pharyngitis streptococcal (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pharyngotonsillitis (Infections and infestations) | 2 (2) | 0 (0) | 1 (1) | 2 (2)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Respiratory tract infection viral (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rhinitis (Infections and infestations) | 3 (3) | 4 (4) | 5 (5) | 7 (7)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Tonsillitis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 2 (2)
Tracheitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tracheobronchitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 8 (8) | 8 (8) | 7 (7) | 4 (4)
Upper respiratory tract infection bacterial (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urethritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 2 (2) | 1 (1) | 2 (2)
Viral infection (Infections and infestations) | 0 (0) | 1 (1) | 3 (3) | 0 (0)
Vulvovaginal mycotic infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Animal bite (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hand fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Joint dislocation (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 54 (55) | 54 (56) | 63 (64) | 34 (36)
Iron deficiency (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 50 (52) | 53 (53) | 49 (55) | 40 (41)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 5 (5) | 4 (4)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 63 (63) | 62 (62) | 58 (63) | 65 (68)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Torticollis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Burning sensation (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (2) | 1 (1) | 1 (1) | 4 (4)
Epilepsy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Generalised tonic-clonic seizure (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 168 (177) | 155 (164) | 178 (200) | 162 (188)
Intercostal neuralgia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Migraine (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Presyncope (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Sciatica (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Tremor (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bulimia nervosa (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Irritability (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypertonic bladder (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dysfunctional uterine bleeding (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dysmenorrhoea (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 1 (1) | 4 (4)
Endometriosis (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Polycystic ovaries (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Adenoidal hypertrophy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 2 (2) | 2 (2)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (2)
Nasal obstruction (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 3 (3) | 1 (1)
Pharyngeal erythema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 3 (3) | 0 (0)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dermal cyst (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hand dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ingrowing nail (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2019-02-08): https://cdn.clinicaltrials.gov/large-docs/82/NCT03433482/Prot_000.pdf
  • Statistical Analysis Plan (2019-07-11): https://cdn.clinicaltrials.gov/large-docs/82/NCT03433482/SAP_001.pdf